CLINICAL TRIAL: NCT00442507
Title: A Phase II Trial of Erlotinib and Avastin in Previously Treated Patients With Cancer of the Esophagus or Gastroesophageal Junction
Brief Title: Erlotinib and Avastin in Patients With Cancer of the Esophagus or Gastroesophageal Junction
Acronym: OSI3650
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-1105
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Results first posted 2015-07-03 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Esophageal Neoplasms; Esophageal Diseases
Keywords: Esophagus; Esophagogastric Junction; Avastin; Bevacizumab; Erlotinib
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Diseases | interventions — Erlotinib Hydrochloride; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients will be treated with erlotinib 150 mg oral daily and Avastin 15 mg/kg intravenously each cycle of therapy (each cycle is 21 days or every 3 weeks). The first infusion of Avastin will be administered over 90 minutes. If tolerated, the second infusion will be given over 60 minutes and in 30 minutes for the subsequent treatments. Treatment will be administered until disease progression or intolerable side effects.
  Interventions: Drug: Erlotinib; Drug: Avastin

INTERVENTIONS:
Drug: Erlotinib
  Other Names: Avastin
Drug: Avastin

SUMMARY:
Determine the time to progression for the combination of erlotinib and bevacizumab in patients with previously treated metastatic cancer of the esophagus or gastroesophageal junction

DETAILED DESCRIPTION:
We postulate that the addition of bevacizumab may increase the efficacy of erlotinib in patients with metastatic esophageal cancer, without adding significant toxicity. The non-overlapping toxicity profiles may allow the administration of the maximum tolerated doses for both agents without additive toxicities with the goal of demonstrating synergistic clinical activity. This combination has been previously tested in two studies for other malignancies with good tolerance and encouraging results.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven adenocarcinoma or squamous cell carcinoma of the esophagus or gastroesophageal junction.
* Metastatic or advanced inoperable disease previously treated with one prior chemotherapy regimen
* Age greater than 18 years.
* Performance status ECOG 0 to 1.
* Adequate hepatic and renal function, defined as:

  * Serum creatinine <= 3.0 mg/dL;
  * Creatinine clearance >= 45 mL/min.
  * Bilirubin <= 1.5 x institutional normal;
  * ALT/AST <= 3 x institutional normal.
* Patients must have measurable disease. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension. The longest diameter of measurable lesions must be >= 20 mm with conventional techniques or >= 10 mm with spiral CT scan. Lesions that are not considered measurable include: bone lesions, leptomeningeal disease, brain lesions, ascites, pericardial or pleural effusion, and tumors situated in a previously irradiated area.
* Use of effective means of contraception for both male and female patients with child-bearing potential.
* A 1 month wash-out period is required for all patients entering this study from a previous treatment regimen

Exclusion Criteria:

* Previous use of anti-EGFR or anti-VEGF therapy.
* Previous history of cancer. The patient with a prior malignancy is eligible for this study only if the patient meets the following criteria for a cancer survivor. A cancer survivor is eligible provided the following criteria are met: (1) patient has undergone potentially curative therapy for all prior malignancies, (2) patients have been considered disease free for at least 5 years (with the exception of basal cell or squamous cell carcinoma of the skin or carcinoma-in-situ of the cervix).
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 0; or anticipation of the need for major surgical procedure during the course of the study. (In the case of high risk procedures such as liver resection, thoracotomy, or neurosurgery, it is recommended that patient delay treatment with chemotherapy for at least 6 weeks and with bevacizumab at least 8 weeks after surgery).
* Radiation therapy within the last 2 weeks.
* Presence of central nervous system or brain metastases at any time.
* Serious, non-healing wound, ulcer, or bone fracture
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to day 0; and/or minor surgical procedures such as fine needle aspiration or core biopsies within 7 days prior to day 0.
* Presence of coagulopathy or clinical history of significant hematemesis, melena, or hemoptysis related to the diagnosis of esophageal cancer.
* Previous history of deep venous thrombosis or thromboembolic disease.
* Urine protein/urine creatinine ratio ≥ 1.0 at screening.
* Pregnant or lactating.
* Unstable angina or history of myocardial infarction within the last 6 months.
* History of stroke within the last 6 months.
* Uncontrolled hypertension with blood pressure persistently > 150/100 mmHg despite optimal antihypertensive therapy.
* Clinically significant peripheral vascular disease.
* Congestive heart failure with New York Heart Association grades III or IV (see appendix B).
* Inability to complete the study and follow-up procedures.
* Participation in therapeutic clinical trials or currently receiving other investigational treatment(s) within 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Morgensztern, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Jemal A, Murray T, Ward E, Samuels A, Tiwari RC, Ghafoor A, Feuer EJ, Thun MJ. Cancer statistics, 2005. CA Cancer J Clin. 2005 Jan-Feb;55(1):10-30. doi: 10.3322/canjclin.55.1.10. PMID 15661684
- [Background] Shah MA, Schwartz GK. Treatment of metastatic esophagus and gastric cancer. Semin Oncol. 2004 Aug;31(4):574-87. doi: 10.1053/j.seminoncol.2004.04.013. PMID 15297948
- [Background] Heath EI, Urba S, Marshall J, Piantadosi S, Forastiere AA. Phase II trial of docetaxel chemotherapy in patients with incurable adenocarcinoma of the esophagus. Invest New Drugs. 2002 Feb;20(1):95-9. doi: 10.1023/a:1014476602804. PMID 12003198
- [Background] Conroy T, Etienne PL, Adenis A, Wagener DJ, Paillot B, Francois E, Bedenne L, Jacob JH, Seitz JF, Bleiberg H, Van Pottelsberghe C, Van Glabbeke M, Delgado FM, Merle S, Wils J. Phase II trial of vinorelbine in metastatic squamous cell esophageal carcinoma. European Organization for Research and Treatment of Cancer Gastrointestinal Treat Cancer Cooperative Group. J Clin Oncol. 1996 Jan;14(1):164-70. doi: 10.1200/JCO.1996.14.1.164. PMID 8558192
- [Background] Lordick F, von Schilling C, Bernhard H, Hennig M, Bredenkamp R, Peschel C. Phase II trial of irinotecan plus docetaxel in cisplatin-pretreated relapsed or refractory oesophageal cancer. Br J Cancer. 2003 Aug 18;89(4):630-3. doi: 10.1038/sj.bjc.6601168. PMID 12915869
- [Background] Mendelsohn J, Baselga J. Status of epidermal growth factor receptor antagonists in the biology and treatment of cancer. J Clin Oncol. 2003 Jul 15;21(14):2787-99. doi: 10.1200/JCO.2003.01.504. PMID 12860957
- [Background] Baselga J, Arteaga CL. Critical update and emerging trends in epidermal growth factor receptor targeting in cancer. J Clin Oncol. 2005 Apr 10;23(11):2445-59. doi: 10.1200/JCO.2005.11.890. Epub 2005 Mar 7. PMID 15753456
- [Background] Johnson JR, Cohen M, Sridhara R, Chen YF, Williams GM, Duan J, Gobburu J, Booth B, Benson K, Leighton J, Hsieh LS, Chidambaram N, Zimmerman P, Pazdur R. Approval summary for erlotinib for treatment of patients with locally advanced or metastatic non-small cell lung cancer after failure of at least one prior chemotherapy regimen. Clin Cancer Res. 2005 Sep 15;11(18):6414-21. doi: 10.1158/1078-0432.CCR-05-0790. PMID 16166415
- [Background] Shepherd FA, Rodrigues Pereira J, Ciuleanu T, Tan EH, Hirsh V, Thongprasert S, Campos D, Maoleekoonpiroj S, Smylie M, Martins R, van Kooten M, Dediu M, Findlay B, Tu D, Johnston D, Bezjak A, Clark G, Santabarbara P, Seymour L; National Cancer Institute of Canada Clinical Trials Group. Erlotinib in previously treated non-small-cell lung cancer. N Engl J Med. 2005 Jul 14;353(2):123-32. doi: 10.1056/NEJMoa050753. PMID 16014882
- [Background] Folkman J. Tumor angiogenesis: therapeutic implications. N Engl J Med. 1971 Nov 18;285(21):1182-6. doi: 10.1056/NEJM197111182852108. No abstract available. PMID 4938153
- [Background] Folkman J. What is the evidence that tumors are angiogenesis dependent? J Natl Cancer Inst. 1990 Jan 3;82(1):4-6. doi: 10.1093/jnci/82.1.4. No abstract available. PMID 1688381
- [Background] Ferrara N, Keyt B. Vascular endothelial growth factor: basic biology and clinical implications. EXS. 1997;79:209-32. doi: 10.1007/978-3-0348-9006-9_9. No abstract available. PMID 9002234
- [Background] Borgstrom P, Gold DP, Hillan KJ, Ferrara N. Importance of VEGF for breast cancer angiogenesis in vivo: implications from intravital microscopy of combination treatments with an anti-VEGF neutralizing monoclonal antibody and doxorubicin. Anticancer Res. 1999 Sep-Oct;19(5B):4203-14. PMID 10628376
- [Background] Presta LG, Chen H, O'Connor SJ, Chisholm V, Meng YG, Krummen L, Winkler M, Ferrara N. Humanization of an anti-vascular endothelial growth factor monoclonal antibody for the therapy of solid tumors and other disorders. Cancer Res. 1997 Oct 15;57(20):4593-9. PMID 9377574
- [Background] Petit AM, Rak J, Hung MC, Rockwell P, Goldstein N, Fendly B, Kerbel RS. Neutralizing antibodies against epidermal growth factor and ErbB-2/neu receptor tyrosine kinases down-regulate vascular endothelial growth factor production by tumor cells in vitro and in vivo: angiogenic implications for signal transduction therapy of solid tumors. Am J Pathol. 1997 Dec;151(6):1523-30. PMID 9403702
- [Background] Hirata A, Ogawa S, Kometani T, Kuwano T, Naito S, Kuwano M, Ono M. ZD1839 (Iressa) induces antiangiogenic effects through inhibition of epidermal growth factor receptor tyrosine kinase. Cancer Res. 2002 May 1;62(9):2554-60. PMID 11980649
- [Background] Ciardiello F, Caputo R, Damiano V, Caputo R, Troiani T, Vitagliano D, Carlomagno F, Veneziani BM, Fontanini G, Bianco AR, Tortora G. Antitumor effects of ZD6474, a small molecule vascular endothelial growth factor receptor tyrosine kinase inhibitor, with additional activity against epidermal growth factor receptor tyrosine kinase. Clin Cancer Res. 2003 Apr;9(4):1546-56. PMID 12684431
- [Background] Jung YD, Mansfield PF, Akagi M, Takeda A, Liu W, Bucana CD, Hicklin DJ, Ellis LM. Effects of combination anti-vascular endothelial growth factor receptor and anti-epidermal growth factor receptor therapies on the growth of gastric cancer in a nude mouse model. Eur J Cancer. 2002 May;38(8):1133-40. doi: 10.1016/s0959-8049(02)00013-8. PMID 12008203
- [Background] Shaheen RM, Ahmad SA, Liu W, Reinmuth N, Jung YD, Tseng WW, Drazan KE, Bucana CD, Hicklin DJ, Ellis LM. Inhibited growth of colon cancer carcinomatosis by antibodies to vascular endothelial and epidermal growth factor receptors. Br J Cancer. 2001 Aug 17;85(4):584-9. doi: 10.1054/bjoc.2001.1936. PMID 11506500
- [Background] Tew WP, Kelsen DP, Ilson DH. Targeted therapies for esophageal cancer. Oncologist. 2005 Sep;10(8):590-601. doi: 10.1634/theoncologist.10-8-590. PMID 16177283
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant accrual on 03/16/2007 and closed to participant accrual on 01/21/2009.
Groups:
- Erlotinib and Avastin: Patients will be treated with erlotinib 150 mg oral daily and Avastin 15 mg/kg intravenously each cycle of therapy (each cycle is 21 days or every 3 weeks). The first infusion of Avastin will be administered over 90 minutes. If tolerated, the second infusion will be given over 60 minutes and in 30 minutes for the subsequent treatments. Treatment will be administered until disease progression or intolerable side effects.
Period: Overall Study
Arm/Group | Erlotinib and Avastin
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib and Avastin
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 63.5 [42 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP)
Description: * TTP is defined as the time from initiation of treatment to the date of documented progression.
  * The median of TTP with 95% confidence interval will be presented.
  * Progressive disease (target lesions) is defined as at least a 20% increase in the sum of the longest diameter of the target lesions taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
  * Progressive disease (non-target lesions) is defined as appearance of one or more new lesions. Unequivocal progression of existing non-target lesions.
Time Frame: Median follow-up for TTP 6 weeks (6-18 weeks)
Population: 1 participant was not analyzed because the participant was removed from study during the first cycle due to an adverse event and was considered not evaluable for this outcome.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib and Avastin
Number analyzed (Participants) | 5
months | 4.2 [1.4 to 13.4]

2. Secondary Outcome: Overall Survival Rate (OS)
Description: OS is defined as the time from initiation of treatment to the date of death for any reason.
Time Frame: Median followup time from completion of treatment 325.5 days (44-401 days)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib and Avastin
Number analyzed (Participants) | 6
months | 10.7 [1.4 to 13.1]

3. Secondary Outcome: Response Rate (Complete Response (CR), Partial Response (PR), and CR+PR)
Description: * CR = disappearance of all target lesions
  * PR = at least a 30% decrease in the sum of the LD of the target lesions taking as reference the baseline sum LD.
Time Frame: Median follow-up for response 6 weeks (6-18 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Erlotinib and Avastin
Number analyzed (Participants) | 5
participants
  Complete response | 0
  Partial response | 0

4. Secondary Outcome: Incidence and Severity of Toxicities
Description: Grade 3 and higher toxicities using CTCAE Version 3.0.
Time Frame: Median follow-up time for toxicities 72 days (72 days-156 days)
Population: Details of all SAEs and AEs are listed in the Serious Adverse Events and Other Adverse Events modules.
Measure: Number; unit: participants
Arm/Group | Erlotinib and Avastin
Number analyzed (Participants) | 6
participants
  Coagulation: Other, IVC Clot | 1
  Death - Disease Progression NOS | 1
  Diarrhea | 1
  GI: Abdominal hemorrhage, NOS | 1
  Pneumonia | 1
  Hypernatremia | 1
  Confusion | 1

ADVERSE EVENTS:
Arm/Group | Erlotinib and Avastin
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib and Avastin (N=6)
Dehydration (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Confusion (Nervous system disorders) | 1
Death - Disease Progression NOS (General disorders) | 1
Coagulation: Other, IVC Clot (Cardiac disorders) | 1
Pneumonia (Infections and infestations) | 1
C. difficile colitis (Infections and infestations) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib and Avastin (N=6)
Atrial flutter (Cardiac disorders) | 1
Hypertension (Vascular disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 2
Sweating (General disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 2
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dyspepsia/heartburn (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Stenosis (Gastrointestinal disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Lymphopenia (Investigations) | 2
Platelets (Investigations) | 1
Bilirubin (Metabolism and nutrition disorders) | 1
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 1
GI: Abdomenal hemorrhage NOS (Gastrointestinal disorders) | 1
Urinary tract infection (Infections and infestations) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 1
Alkaline phosphatase (Metabolism and nutrition disorders) | 2
Confusion (Nervous system disorders) | 1
Cerebrovascular ischemia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Mood alteration - depression (Psychiatric disorders) | 1
Neuropathy (Nervous system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Chest pain (Cardiac disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Limb pain (Musculoskeletal and connective tissue disorders) | 1
Esophagus pain (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine (Investigations) | 1
Hematuria (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes